CLINICAL TRIAL: NCT03965156
Title: Bilateral Ultrasound Guided Erector Spinae Plane Block Versus Transversus Abdominis Plane Block on Post-operative Analgesia After Total Abdominal Hysterectomy
Brief Title: Bilateral Ultrasound Guided ESP Block Versus TAP Block on Post-operative Analgesia After Total Abdominal Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Alshaimaa Abdel Fattah Kamel, lecturer of Anaesthesia ,and surgical intensive care, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5423
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Post-operative Analgesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spinae Plane Block (Active Comparator): Bilateral Ultrasound Guided Erector Spinae Plane Block
  Interventions: Procedure: 1) Ultrasound guided Erector spinae block
- transversus abdominis plane block (Active Comparator): Ultrasound guided transversus abdominis plane block
  Interventions: Procedure: Ultrasound guided transversus abdominis plane block

INTERVENTIONS:
Procedure: 1) Ultrasound guided Erector spinae block — In the lateral position, after skin sterilization, erector spinae plane block will be performed at the level of T9. Counting down from the spine of seventh cervical vertebrae, the spine of the nine thoracic vertebrae (T9). A linear low frequency ultrasound transducer (US) (3-5 MHz) will placed sagittal 3cm lateral to midline to visualize the muscles of the back, transverse process and simmering pleura in between transverse processes. A 22-gauge short bevel needle will be inserted in cranial-caudal direction towards transverse process (TP) in plane to the US transducer until needle touched the TP crossing all the muscles. The location of the needle tip will be confirmed by visible normal saline fluid separating erector spinae muscle off the bony shadow of the transverse process on ultrasound imaging. Then 20 ml of bupivacaine 0.375% plus plus 5ug/ml adrenaline (1:200000) will be injected. The procedure will be repeated following the same steps on the other side of the back.
  Arms: Erector Spinae Plane Block
Procedure: Ultrasound guided transversus abdominis plane block — in supine position and after skin sterilization. The linear high frequency transducer (6-13 MHz) will be placed in the transverse plane to the the lateral abdominal wall in the midaxillary line, between the lower costal margin and iliac crest. The three abdominal wall muscles (external oblique, internal oblique, and transversus abdominis) are visualized. The needle inserted in plane and advanced anterior to posterior under continual visualization until the tip between the internal oblique and the transversus abdominis muscle. After negative aspiration, a 20 ml of bupivacaine 0.375% plus 5ug/ml adrenaline (1:200000) will be injected. The success of the injection will be confirmed by separation of the internal oblique and transversus abdominis with a distinct pocket of local anesthetic in between. The procedure will be repeated following the same steps on the other side.
  Arms: transversus abdominis plane block

SUMMARY:
* Abdominal hysterectomy is an open surgical procedure associated with considerable post-operative pain. Narcotics are often required during patient recovery but can result in adverse side effects. Transversus abdominis plane block(TAP block) is a regional anesthetic technique that is found to be effective as post-operative analgesia after total abdominal hysterectomy. Recently, erector spinae plane block(ESP)block is found to be safe, and simple regional anesthetic technique that decrease total opioid consumption in patient undergoing breast, or abdominal surgery.
* The aim is to compare the efficacy of bilateral erector spinae plane block, and bilateral transversus abdominis plane block on postoperative analgesia in patients after abdominal hysterectomy under general anesthesia, and their need for opioid.

Hypothesis

* Null hypothesis (H0): No difference between the analgesic effects of bilateral erector spinae plane block, and bilateral transversus abdominis plane block in patients after abdominal hysterectomy under general anesthesia.
* Alternative hypothesis (H1): There are difference between the analgesic effects of bilateral erector spinae plane block, and bilateral transversus abdominis plane block in patients after abdominal hysterectomy under general anesthesia.

DETAILED DESCRIPTION:
Sample size: Assuming that Mean±SD of reduced pain scores in erector spinae plane block is 4.7±3.7 versus 2.5±1 in transversus abdominis plane block.So, the total sample size is 48 cases (24 in each group) using Open Source Statistics for Public Health (open Epi) with confidence interval 95% and power of test is 80%.

d) Method of sample collection:

Forty eight female patients will be divided into two groups by a computer-generated randomization table:

Group (ES) (n=24): will receive bilateral ultrasound guided erector spinae plane block with each block 20 ml of bupivacaine 0.375% plus 5ug/ml adrenaline (1:200000) at the level of T9.

Group (TA) (n=24): will receive bilateral ultrasound guided transversus abdominis plane block with each block 20 ml of bupivacaine 0.375% plus 5ug/ml adrenaline (1:200000).

ELIGIBILITY:
Inclusion Criteria:

* Female Patient.
* Patient acceptance.
* Age (40-60) years old.
* American Society of Anaesthesiologist (ASA) I / II
* Elective total abdominal hysterectomy under general anesthesia.
* patient With Body Mass Index (BMI) (25-35kg/m²)

Exclusion Criteria:

* Patient refusal.
* Local infection at site of puncture.
* Altered mental status.
* History of allergy to study drugs ( bupivacaine, morphine).
* Patients with chronic pain.
* Patients with severe hepatic or kidney impairment.
* Patients having a history of hematological disorders, including coagulation abnormality.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-11 (Actual)

PRIMARY OUTCOMES:
The total amount of morphine given to each patient | the first 24 hours postoperative.
  The total amount of morphine given to each patient during the first 24h of postoperative period
The time to first call to analgesia (morphine) | first call to morphine up to 24 hours postoperative.
  morphine (rescue analgesic) will be given if VAS>3.
Pain intensity using Visual analogue Scale (VAS) (McCormack et al., 1988). | at 30 minutes postoperative.
  1- Pain intensity using Visual analogue Scale (VAS) (McCormack et al., 1988). A commonly used visual analog scale is a 10-cm line labeled with "worst pain imaginable" on the right border and "no pain" on the left border. The patient is instructed to make a mark along the line to represent the intensity of pain currently being experienced. VAS score will be assessed at 30 minutes, 2hs, 4hs, 6hs, 12hs, and 24hs postoperative and IV increment of 3mg morphine (rescue analgesic) will be given if VAS>3.
Pain intensity using Visual analogue Scale (VAS) | at 2 hours postoperative.
  visual analogue scale is a 10-cm line labeled with "worst pain imaginable" on the right border and "no pain" on the left border.
Pain intensity using Visual analogue Scale (VAS) | at 4 hours postoperative.
  visual analogue scale is a 10-cm line labeled with "worst pain imaginable" on the right border and "no pain" on the left border.
Pain intensity using Visual analogue Scale (VAS) | at 6 hours postoperative.
  visual analogue scale is a 10-cm line labeled with "worst pain imaginable" on the right border and "no pain" on the left border.
Pain intensity using Visual analogue Scale (VAS) | at 12 hours postoperative.
  visual analogue scale is a 10-cm line labeled with "worst pain imaginable" on the right border and "no pain" on the left border.
Pain intensity using Visual analogue Scale (VAS) | at 24 hours postoperative.
  visual analogue scale is a 10-cm line labeled with "worst pain imaginable" on the right border and "no pain" on the left border.
"Number of Participants with nausea, Vomiting, nausea or vomiting, hypotension, bradycardia, or any other complication" | Up to 24 hours postoperative.
  "Number of Participants with nausea, Vomiting, nausea or vomiting, hypotension, bradycardia, or any other complication"

SECONDARY OUTCOMES:
Over all patient satisfaction | all over 24 hours postoperative
  Over all patient satisfaction:The patients will be asked to rate the overall degree of satisfaction of the analgesia using a 1-3 verbal scale (1 = unsatisfactory analgesia, 2 = satisfactory analgesia, and 3 = excellent analgesia) (Ross et al., 2009).

CONTACTS AND LOCATIONS:
Overall Officials: Alshaimaa Kamel, M.D, Principal Investigator — faculty of medicine ,zagazig universty
Locations (1):
- Zagazig University Hospitsals, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No